CLINICAL TRIAL: NCT02299271
Title: Fascia Iliaca Block for Post-Operative Pain Control After Total Hip Arthroplasty: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Fascia Iliaca Block for Post-Operative Pain Control After Total Hip Arthroplasty
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Preliminary analysis showed no difference between groups.
Sponsor: The Christ Hospital (Other)
Responsible Party: Principal Investigator, Brian Vaughan, Brian Vaughan, MD, The Christ Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Christh-01
Record Dates: First submitted 2014-11-19; First posted 2014-11-24 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Osteoarthritis of the Hip
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ropivacaine block (Active Comparator): Ropivacaine 0.375% as a one-time 60 milliliter injection.
  Interventions: Drug: Ropivacaine
- saline block (Placebo Comparator): Sodium chloride 0.9% as a one-time 60 milliliter injection.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine — 0.375% ropivacaine as a one-time, 60 milliliter injection
  Other Names: Naropin
  Arms: ropivacaine block
Drug: Saline — Saline as a one-time, 60 milliliter injection.
  Other Names: Sodium Chloride 0.9%
  Arms: saline block

SUMMARY:
This study evaluates post-operative pain management and narcotic consumption in patients receiving a fascia iliaca block with local anesthetic versus patients receiving fascia iliaca block with saline for total hip arthroplasty.

DETAILED DESCRIPTION:
Although many improvements have been made in implant technology and surgical approaches for total hip arthroplasty, management of post-operative pain remains a major clinical issue. Inadequate pain control can lead to numerous unwanted side effects and limited physical function, especially in a older population. Most surgeons have adopted a multi-modality pain management approach using a variety of pharmaceuticals, including nerve block with local anesthetic. In the literature, there are a number of technical variations described for the fascia iliaca nerve block. At The Christ Hospital, Cincinnati, Ohio, anesthesiologists use a more proximal approach to the fasica iliaca block enabling a significantly easier cephalad spread of the local anesthetic into the pelvis targeting all three nerves; the femoral, lateral femoral cutaneous, and the obturator.

This prospective, double-blinded, randomized, single-center study is designed to test the primary hypothesis that fascia iliaca block with a local anesthestic decreases narcotic consumption and provides improved pain control compared to placebo in the first 24 hours after surgery in patients undergoing total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* anterior approach total hip arthroplasty (THA) for unilateral osteoarthritis
* English-speaking
* age 18 to 75 years
* American Society of Anesthesiologists (ASA) physical status 1 to 3
* BMI < 40 kg/m2
* Minimum weight of 50 kg.
* No contraindications to study procedures

Exclusion Criteria:

* Hip revision surgery
* Allergy to local anesthetics
* Allergy to oxycontin
* Allergy to pregabalin
* Allergy to fentanyl
* Allergy to midazolam
* Allergy to hydromorphone
* BMI > 40 kg/m2
* Chronic pre-operative opioid use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain Control | 24 hours
  Measured by NRS-11 beginning in post-operative care unit and continuing 24 hours on the post-operative floor.
Opioid Consumption | 24 hours
  Measured by IV narcotic consumption beginning in the post-operative care unit and continuing 24 hours on the post-operative floor.

SECONDARY OUTCOMES:
Post-Operative Care Unit (PACU) Length of Stay | From 60 minutes to 6 hours
  Length of PACU stay is measured from arrival in PACU to clinical discharge from PACU

CONTACTS AND LOCATIONS:
Overall Officials: Brian Vaughan, MD, Principal Investigator — The Christ Hospital
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Shariat AN, Hadzic A, Xu D, Shastri U, Kwofie K, Gandhi K, McCally CM, Gratenstein K, Vandepitte C, Gadsden J, Unis D. Fascia lliaca block for analgesia after hip arthroplasty: a randomized double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2013 May-Jun;38(3):201-5. doi: 10.1097/AAP.0b013e31828a3c7c. PMID 23558369